CLINICAL TRIAL: NCT01957904
Title: Prospective, Multi-Center, Open-Label, Post-Market ArterX® Safety and Efficacy Study Protocol for Cardiac Indications
Brief Title: ArterX Safety and Efficacy Study for Cardiac Indications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tenaxis Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN-015
Record Dates: First submitted 2013-09-27; First posted 2013-10-08 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Vascular Disease
Keywords: ArterX, surgical sealant
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ArterX Surgical Sealant (Other)
  Interventions: Device: ArterX Surgical Sealant

INTERVENTIONS:
Device: ArterX Surgical Sealant

SUMMARY:
The study is designed to confirm the acute safety and performance of the ArterX® Surgical Sealant as a hemostatic agent. The study will collect data in support of publications and future product labeling revisions, to provide additional clinical information on use and further details regarding product safety.

ELIGIBILITY:
Inclusion Criteria:

>18 years of age, Male or female If female, subject is post-menopausal, has no child bearing potential or has a negative serum or urine pregnancy test within 7 days of the index procedure and is practicing abstinence or a highly effective method of contraception for the duration of the study.

The subject or guardian must provide written Informed Consent using a form that is reviewed and approved by the Ethics Committee.

The subject is willing and able to be contacted for 3 months follow-up and attend follow-up visits as needed per protocol.

The subject is determined by the surgeon to be at risk for poor hemostasis.

Exclusion Criteria:

Subject undergoing emergency surgery. Subject undergoing minimally invasive surgery. Subject has clinically significant medical, psychiatric, or cognitive illness or drug/alcohol abuse that in the opinion of the investigator would affect the subject's safety or compliance with study assessments or follow-up.

Subject has immune system disorders/immunodeficiency or immunosuppression. Subject has participated in another clinical study within 30 days prior to surgery or has received an investigational drug or device within the past 30 days.

Subject is pregnant, may become pregnant or is currently breast feeding

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects with immediate sealing of suture/staple line | during surgery
  Immediate sealing of the suture/staple line at point of use upon release of the clamps, as evidenced by an absence of clinically significant bleeding as determined by physician investigator in procedures completed using the ArterX device.

CONTACTS AND LOCATIONS:
Locations (1):
- Krankenhaus Der Barmherzigen Bruder, Trier, Germany

REFERENCES:
- [Result] Skorpil J, Paraforos A, Mandak J, Cohn WE, Hajek T, Friedrich I. Effective and rapid sealing of coronary, aortic and atrial suture lines dagger. Interact Cardiovasc Thorac Surg. 2015 Jun;20(6):720-4; discussion 724. doi: 10.1093/icvts/ivv061. Epub 2015 Mar 24. PMID 25810290